CLINICAL TRIAL: NCT06154278
Title: Pilot Study to Evaluate Intrahepatic and Peripheral Responses to Small Interfering RNA, Imdusiran (AB-729), Among People With Chronic Hepatitis B
Brief Title: Intrahepatic and Peripheral Responses to Imdusiran (AB-729) in Chronic Hepatitis B
Acronym: i-LIVER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Arbutus Biopharma Corporation (Industry)
Responsible Party: Principal Investigator, Lydia Tang, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00106061
Record Dates: First submitted 2023-10-31; First posted 2023-12-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
Keywords: hepatitis B; SiRNA; liver biopsy; Imdusiran
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, pilot study of Imdusiran (AB-729) in virally suppressed adults with chronic hepatitis B on oral antiviral therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imdusiran (AB-729) (Experimental): Participants receive subcutaneous injections of 60mg, one injection every 8 weeks for 4 doses.
  Interventions: Drug: Imdusiran (AB-729)

INTERVENTIONS:
Drug: Imdusiran (AB-729) — 60mg subcutaneously, every 8 weeks, for a total of 4 doses

SUMMARY:
The goal of this clinical trial is to learn about the action of Imdusiran (AB-729) in the liver of people with chronic hepatitis B. The main questions it aims to answer are:

* how well is it working in the liver
* how does Imdusiran affect the hepatitis B virus

Participants will receive injections of Imdusiran, one injection every 8 weeks, for a total of 4 doses. They will also undergo 2 liver biopsies: one with the first dose of Imdusiran, and the second 8 weeks after the last dose of Imdusiran.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, pilot study of Imdusiran in adults with chronic hepatitis B on oral antiviral therapy. The primary objective of this study is to evaluate the intrahepatic concentrations of Imdusiran. The secondary objective is to evaluate the effect of Imdusiran on viral markers.

Up to 10 participants will receive a total of 4 subcutaneous injections of 60mg Imdusiran (one injection every 8 weeks). They will undergo 2 liver biopsies: one with the first dose, and the second 8 weeks after the last dose. There is an optional third liver biopsy at the end of study (week 52).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, over 18 years of age on the date of screening
4. In good general health as evidenced by medical history
5. Documented evidence of chronic hepatitis B infection (HBsAg positive at screening and for at least more than 6 months prior to screening)
6. For females of reproductive potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline prior to study drug administration
7. Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
8. Have been on commercially available HBV oral antiviral treatment(s) for at least 6 months and willing to continue through the final study visit.
9. HBV Deoxyribonucleic acid (DNA) ≤ 20 IU/mL for 6 or more months prior to Screening.
10. Hepatitis B surface antigen titer ≥ 100 IU/mL.
11. Liver imaging without liver mass suggestive of hepatocellular carcinoma within 12 months of day 0 AND Alpha fetoprotein <10 ng/mL within 3 months of screening.

Exclusion Criteria:

1. Known co-infection with any of the following:

   1. Human immunodeficiency virus (HIV)
   2. Hepatitis C virus (HCV), unless subjects are HCV Ab positive, but have a documented history of completing HCV treatment and/or negative HCV RNA
   3. Hepatitis D virus (HDV)
2. Any known preexisting medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study
3. History of cirrhosis at any time, or evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding esophageal varices, hepatorenal syndrome, liver transplantation and/or hepatic encephalopathy.
4. Liver ultrasound or other imaging with findings suggestive of hepatocellular carcinoma (HCC) at any time.
5. Clinically unstable medical condition ≤2 weeks prior to the first dose of study treatment.
6. Clinical diagnosis of substance abuse with alcohol, narcotics, or cocaine within the past 12 months except for those subjects monitored in an opioid substitution maintenance program.
7. Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (e.g. basal cell skin cancer). Subjects under evaluation for possible malignancy are not eligible.
8. Extensive bridging fibrosis or cirrhosis as defined clinically, by imaging or by the following:

   a. Metavir ≥ 3 or Ishak fibrosis score ≥ 4 by a liver biopsy within 3 years of screening, or, in the absence of an appropriate liver biopsy, either: i. Screening FibroTest score >0.48 and APRI >1, or ii. FibroScan with a result >9 kPa within 12 months of screening
   * If liver biopsy is available, the liver biopsy result supersedes (i) and (ii).
9. Subjects meeting any of the following laboratory parameters at screening:

   1. Alanine aminotransferase (ALT) >3x Upper Limit of Normal (ULN)
   2. Direct bilirubin (if total bilirubin elevated) >1.5 × ULN of the laboratory reference range.
   3. Prothrombin (PT) or Activated Partial Thromboplastin Clotting Time (APTT) over the upper limit of normal.
   4. Platelet count <100,000/microliters
   5. Estimated glomerular filtration rate, calculated by the chronic kidney disease epidemiology collaboration formula: <60 mL/min/1.73 m2
10. Significant cardiovascular, pulmonary, or neurological disease in the opinion of the investigator.
11. Participation in any investigational drug, vaccine, or device study within 30 days before study treatment administration, or 90 days for a biologic study, or at any time during participation in the study.
12. Pregnancy or lactation
13. Believed by the Study Investigator to be inappropriate for study participation for any reason not otherwise listed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic concentration of Imdusiran (AB-729) | During intervention (with first dose of Imdusiran) and after intervention (8 weeks after last dose of Imdusiran)
  Intrahepatic drug concentration at day 0 (peak) and week 32 (trough)

SECONDARY OUTCOMES:
Effect of Imdusiran (AB-729) on hepatitis B surface antigen production | Baseline through study completion, an average of 1 year
  Change in hepatitis B surface antigen titer with Imdusiran
Effect of Imdusiran (AB-729) on hepatitis B surface antibody levels | Baseline through study completion, an average of 1 year
  Change in hepatitis B surface antigen-specific antibody levels (anti-HBsAg)
Effect of Imdusiran (AB-729) on hepatitis B virus RNA | Baseline through study completion, an average of 1 year
  Change in HBV RNA production
Effect of Imdusiran (AB-729) on hepatitis B virus e antigen production | Baseline through study completion, an average of 1 year
  Change in quantitative HBeAg
Effect of Imdusiran (AB-729) on hepatitis B surface antigen serostatus | Baseline through study completion, an average of 1 year
  Proportion of participants with hepatitis B surface antigen loss
Effect of Imdusiran (AB-729) on hepatitis B surface antibody serostatus | Baseline through study completion, an average of 1 year
  Proportion of participants with anti-HBsAg seroconversion
Effect of Imdusiran (AB-729) on hepatitis B e antigen serostatus | Baseline through study completion, an average of 1 year
  Proportion of participants with HBeAg loss
Effect of Imdusiran (AB-729) on hepatitis B e antibody serostatus | Baseline through study completion, an average of 1 year
  Proportion of participants with anti-HBeAg seroconversion

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Human Virology, University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No